CLINICAL TRIAL: NCT06198296
Title: Immunotherapy For Adults With GPC3-Positive Solid Tumors Using Interleukin-15 And -21 Armored Glypican-3-Specific Chimeric Antigen Receptor Expressing Autologous T Cells
Brief Title: Immunotherapy For Adults With GPC3-Positive Solid Tumors Using IL-15 and IL-21 Armored GPC3-CAR T Cells
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Premal Lulla, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-54859 CO-EXIST
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Hepatoblastoma; Hepatocellular Carcinoma; Wilms Tumor; Malignant Rhabdoid Tumor; Yolk Sac Tumor; Rhabdomyosarcoma; Liposarcoma; Embryonal Sarcoma of Liver
Keywords: GPC3-positive tumors; GPC3-CAR T cells
MeSH Terms: conditions — Hepatoblastoma; Carcinoma, Hepatocellular; Wilms Tumor; Rhabdoid Tumor; Endodermal Sinus Tumor; Rhabdomyosarcoma; Liposarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 21.15.GPC3-CAR T cells (Experimental): GPC3-CAR and the IL15 plus IL21 will be administered to patients with GPC3-positive solid tumors.
  Interventions: Genetic: 21.15.GPC3-CAR T cells

INTERVENTIONS:
Genetic: 21.15.GPC3-CAR T cells — Three different dosing schedules will be evaluated.
  The following dose levels will be evaluated:
  The following dose levels will be evaluated:
  DL0: 3x10^7/m2 DL1: 1x10^8/m2 DL2: 3x10^8/m2 DL3: 1x10^9/m2

SUMMARY:
The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancers. This research study combines two different ways of fighting cancer: antibodies and T cells.

Antibodies are types of proteins that protect the body from infectious diseases and possibly cancer. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including cells infected with viruses and tumor cells. Both antibodies and T cells have been used to treat patients with cancers. They have shown promise but have not been strong enough to cure most patients.

In order to get them to kill cancers more effectively, in the laboratory, the study team inserted a new gene called a chimeric antigen receptor (CAR) into T cells that makes them recognize cancer cells and kill them. When inserted, this new CAR T cell can specifically recognize a protein found on solid tumors, called glypican-3 (GPC3). To make this GPC3-CAR more effective, the study team also added two genes called IL15 and IL21 that help CAR T cells grow better and stay in the blood longer so that they may kill tumors better. When the study team did this in the laboratory, they found that this mixture of GPC3-CAR,IL15 and IL21 killed tumor cells better when compared with CAR T cells that did not have IL15 plus IL21 in the laboratory. This study will use those cells, which are called 21.15.GPC3-CAR T cells, to treat patients with solid tumors that have GPC3 on their surface.

The study team also wanted to make sure that they could stop the 21.15.GPC3-CAR T cells from growing in the blood should there be any bad side effects. In order to do so, they inserted a gene called iCasp9 into the CO-EXIST T cells. This allows us the elimination of 21.15.GPC3-CAR T cells in the blood when the gene comes into contact with a medication called AP1903. The drug (AP1903) is an experimental drug that has been tested in humans with no bad side-effects. This drug will only be used to kill the T cells if necessary due to side effects .

The study team has treated patients with T cells that include GPC3. Patients have also been treated with IL-21 and with IL-15. Patients have not been treated with a combination of T cells that contain GPC3, IL-21 and IL-15. To summarize, this study will test the effect of 21.15.GPC3-CAR T cells in patients with solid tumors that express GPC3 on their surface.

The 21.15.GPC3-CAR T cells are an investigational product not yet approved by the Food and Drug Administration.

DETAILED DESCRIPTION:
The study team will collect up to 18 teaspoons of patients' blood. This will be used this blood to grow T cells. The study team then grows the T cells and uses a retrovirus (a special virus that can insert the GPC3 CAR and IL15 plus IL21 genes into the T cells) to genetically engineer (generate cells in the laboratory) them. After the CAR and IL15 plus IL21 genes are put into the T cells, the study team ensures that they could kill GPC3 positive solid tumor cells in the laboratory.

LYMPHODEPLETION CHEMOTHERAPY:

Several studies suggest that the infused T cells need room to be able to proliferate and accomplish their functions and that this may not happen if there are too many other T cells in the blood . Lymphodepletion chemotherapy is a way of temporarily decreasing the amount of the body s T cells , so that CO-EXIST T cells can grow better. with the two lymphodepleting chemotherapy drugs we will use are called cyclophosphamide (Cytoxan) and fludarabine. They will both be given daily for 3 days before receiving the T-cell infusion.

WHAT THE INFUSION WILL BE LIKE:

If you agree to participate in this study, at the time you are scheduled to be treated, the cells will be thawed and injected into you over 5 to 10 minutes. You will receive the CO-EXIST T cells 48 to 72 hours after completing the chemotherapy. You may be given Tylenol (acetaminophen) and Benadryl (diphenhydramine) before the CO-EXIST T cells to prevent a possible allergic reaction.

This is a dose escalation study, which means that the study team does now know the highest dose of 21.15.GPC3-CAR T cells that is safe. To find out, the cells will be given to at least 3 participants at a lower dose. If that is safe, the study team will raise the dose level that is given to the next group of participants. The dose a patient received will get will depend on how many participants get the agent before the patient and how they react. The investigator will tell the patient this information. Since the treatment is experimental, what is likely to happen at any dose is not known.

If after 4 weeks the patient's condition does not get worse, the patient may receive another round of lymphodepleting chemotherapy and infusion of 21.15.GPC3-CAR T cells.

All the treatments will be given by the Center for Cell and Gene Therapy at Methodist Hospital of Houston.

Medical tests before treatment:

Before being treated, the patient will receive a series of standard medical tests:

* Physical exam and history
* Blood tests to measure blood cells, kidney and liver function.
* Pregnancy test (if the patient is a female who can get pregnant)
* If the patient is infected with the hepatitis B virus (HBV) sthe study team will do a test to measure the levels of the virus
* Measurements of the patient's tumor by scans (either CT or MRI). Side effects are rare and include risk of developing an unrelated cancer due to radiation exposure from the machine, but this is unlikely.
* the tumor marker alfa-fetoprotein (AFP), if the patient's tumor produces this protein.

Medical tests during and after treatment:

The patient will receive standard medical tests when you are getting the infusions and after:

* Physical exams and History
* Blood tests to measure blood cells, kidney and liver function.
* If the patient is infected with the hepatitis B virus (HBV) the study team will repeat the test and monitor the levels of the virus
* Measurements of the patient's tumor by scans (same scans used before treatment) (4 - 6 weeks after the infusion) and AFP (if applicable at 1, 2, and 4 weeks after the infusion).
* Tumor biopsy of an accessible tumor between 2-4 weeks after the infusion and as clinically indicated thereafter. For additional clinically indicated tumor biopsies the study team will ask for a portion of the sample for research. The study team will not obtain biopsies if the patient's tumors are not accessible.

FOLLOW-UP STUDIES:

The study team will follow the patient during and after the injections. To learn more about the way the T cells are working in the patient's body, up to 60 mL (up to 12 teaspoons) of blood will be taken from the patient before the chemotherapy, before the T-cell infusion, 1 to 4 hours after the infusion, 3 to 4 days after the infusion (this time point is optional ) at 1 week, 2 weeks, 4 weeks and 8 weeks after the injection, every 3 months for 1 year, every 6 months for 4 years and then every year for the next 10 years. Total participation time for this study will be 15 years.

During the time points listed above, if the T cells are found in the patient's blood at a certain amount an extra 5mL of blood may need to be collected for additional testing .

The study team will use this blood to look for the frequency and activity of the cells that we have given; that is, to learn more about the way the T cells are working and how long they last in the body. The study team will also use this blood to see if there are any long-term side effects of putting the new gene (chimeric antigen receptor, CAR) into the cells. In addition to the blood draws, because the patient will receive cells that have had a new gene put in them, the patient will need to have long term follow up for 15 years so the study team can see if there are any long-term side effects of the gene transfer.

Once a year, the patient will be asked to have blood drawn and answer questions about their general health and medical condition. The investigators may ask the patient to report any recent hospitalizations, new medications, or the development of conditions or illness that were not present when the patient enrolled in the study and may request that physical exams and/or laboratory tests be performed if necessary.

When tumor biopsy is performed for clinical reasons the study team will request permission to obtain excess sample to learn more about the effects of the treatment on the patient's disease.

In the event of death, the study team will request permission to perform an autopsy (a procedure where a doctor examines the body to look for a cause of death) to learn more about the effects of the treatment on the patient's disease and if there were any side effects from the cells with the new gene.

In addition, the study team will ask for your permission to use tumor biopsy for research purposes only. Associated risk with the biopsy will be discussed with the patient in detail in a procedure specific consent form. The study team will test the sample to see if the 21.15.GPC3-CAR T cells can be found in the tumor and what effect they had on the tumor cells.

If the patient develops a second abnormal cancer growth, significant blood or nervous system disorder during the trial, the study team will request that a biopsy sample of the tissue will be tested.

The remaining blood and/or tissue samples that are not needed directly for the patient could be used to help researchers learn about this disease and/or immune therapy. These specimens and information about the patient's circumstances may be shared with other cancer researchers. Although there will be a record identifying under what circumstances these specimens were obtained, under all circumstances the patient's identity will be kept confidential. There is a small risk for the loss of confidentiality. However, study personnel will make every effort to minimize this risk. Samples will be kept at Baylor College of Medicine until they are exhausted.

ELIGIBILITY:
Procurement Inclusion Criteria:

* Diagnosis of GPC3-positive* solid tumors (as determined by immunohistochemistry with an extent score of >=Grade 2 [>25% positive tumor cells] and an intensity score of >= 2 [scale 0-4]).
* Age ≥21 years
* Lansky or Karnofsky score ≥60%
* Life expectancy ≥16 weeks
* Barcelona Clinic Liver Cancer Stage A, B or C (- Child-Pugh-Turcotte score <7 (for patients with hepatocellular carcinoma only)
* Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent * GPC3 expression will be evaluated by standard immunohistochemistry (IHC) at Texas Patients's Hospital/Baylor College of Medicine, Department of Pathology for all patients to meet procurement eligibility. All patients will send at least 5 unstained slides.

Procurement Exclusion Criteria:

* History of hypersensitivity reactions to murine protein-containing products OR presence of human anti-mouse antibody (HAMA) prior to enrollment (only patients who have received prior therapy with murine antibodies).
* History of organ transplantation
* Known HIV positivity
* Active bacterial, fungal or viral infection (except Hepatitis B or Hepatitis C virus infections)

Treatment Inclusion Criteria:

* Diagnosis of GPC3-positive solid tumor
* Age ≥ 21 years
* Barcelona Clinic Liver Cancer Stage A, B or C
* Life expectancy of ≥ 12 weeks
* Lansky or Karnofsky score ≥ 60%
* Child-Pugh-Turcotte score < 7
* Adequate organ function:
* Creatinine clearance as estimated by Cockcroft Gault or Schwartz ≥ 60 ml/min
* total bilirubin < 3 times ULN for age
* INR ≤1.7 (for patients with hepatocellular carcinoma only)
* absolute neutrophil count > 500/µl
* platelet count > 25,000/µl (can be transfused)
* Hgb ≥ 7.0 g/dl (can be transfused)
* Pulse oximetry >90% on room air
* Refractory or relapsed disease after treatment with up- front therapy and at least one salvage treatment cycle
* Recovered from acute toxic effects of all prior chemotherapy and investigational agents before entering this study, as determined by history and physical exam
* Sexually active patients must be willing to utilize one of the more effective birth control methods for 3 months after the T-cell infusion.
* Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent

Treatment Exclusion Criteria:

* Pregnancy or lactation
* Uncontrolled infection
* Systemic steroid treatment (greater than or equal to 0.5 mg prednisone equivalent/kg/day, dose adjustment or discontinuation of medication must occur at least 24hrs prior to CAR T cell infusion)
* Known HIV positivity
* Active bacterial, fungal or viral infection (except Hepatitis B or Hepatitis C virus infections)
* History of organ transplantation
* History of hypersensitivity reactions to murine protein-containing products OR presence of human anti-mouse antibody (HAMA) prior to enrollment (only patients who have received prior therapy with murine antibodies)

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2043-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose Limiting Toxicity | 4 weeks
  A dose limiting toxicity is defined as any toxicity that is considered to be primarily related to the GPC3-CAR T cells. Specifically those which are Grade 5; non-hematologic Grade 3-4 not returning to Grade 2 within 72 hours; Grade 2-4 allergic reaction; Hematologic Grade 4 that fails to return to Grade 2 or baseline (whichever is more severe) within 14 days; all grade 4 CRS and neurologic toxicities and grade 3 CRS and neurologic toxicities that fail to return to Grade 1 within 7 days

SECONDARY OUTCOMES:
Percent of Patients with best response as either complete remission or partial remission | 4 weeks
  Response rates will be estimated as the percent of patients whose best response is either complete remission or partial remission by combining the data from the two patients. To compare with historical data, a 95% confidence interval will be calculated for the response rate
Median T cell persistence | 15 years
  T cell persistence will be measured by PCR

CONTACTS AND LOCATIONS:
Overall Officials: Premal Lulla, MD, Principal Investigator — Baylor College of Medicine; David Steffin, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States